CLINICAL TRIAL: NCT05468151
Title: Cold Acclimation As a Modulator of Brown Adipose Tissue Function in Adults with Obesity
Acronym: MOTORBAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); University of Barcelona (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Kirsi Virtanen, Associate Professor at Turku PET Centre, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T138/2022
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cold acclimation protocol (Experimental): Participants with obesity (n = 20) will undergo weekly cold water immersions (water temperature 18ºC, two to three times a week, 30 minutes per day) for, at least, 12 weeks. Before and after the cold acclimation period, the participants will undergo PET/CT scans at room temperature and after controlled cold exposure to investigate BAT perfusion, BAT glucose and NEFA uptakes.
  Interventions: Other: Cold acclimation
- Acute cold exposure - control volunteers with obesity (Other): PET/CT scans will be carried out after 2 hours of cold exposure The participants in this group (n = 10) will undergo PET/CT scans at baseline and 12 weeks after the first scan.
  The participants will undergo PET/CT scans at room temperature and after 2 hours of controlled cold exposure to investigate BAT perfusion, BAT glucose and NEFA uptakes.
  Interventions: Other: Intervention Control group - volunteers with obesity
- Acute cold exposure - lean controls (Other): PET/CT scans will be carried out after 2 hours of cold exposure The participants in this group (lean, n = 15) will undergo PET/CT scans at room temperature and after 2 hours of controlled cold exposure to investigate BAT perfusion, BAT glucose and NEFA uptakes.
  Interventions: Other: Acute cold exposure

INTERVENTIONS:
Other: Cold acclimation — The cold water immersions will last 30-60 minutes per day and the volunteers will undergo 2-3 cold immersions per week.
  Other Names: Cold immersion
  Arms: Cold acclimation protocol
Other: Intervention Control group - volunteers with obesity — Participants with obesity in the control group will undergo PET/CT scans at baseline and 12 weeks after the first scan.
  Arms: Acute cold exposure - control volunteers with obesity
Other: Acute cold exposure — All participants (lean and with obesity) will undergo PET/scans after 2 hours of cold exposure to investigate BAT perfusion and BAT glucose uptake.
  Arms: Acute cold exposure - lean controls

SUMMARY:
This study will investigate the effects of at least 12 weeks of weekly cold water immersions (water temperature 18ºC) on BAT perfusion in individuals with obesity. BAT oxygen uptake and tissue perfusion will be measured using 15O-O2 and 15O-H2O PET-CT, at room temperature and after cold exposure. In addition, BAT glucose uptake will be measured using 18F-FDG after 2 hours of cold exposure and BAT NEFA uptake will be analyzed using 18F-FTHA at room temperature.

To understrand the metabolic effects of BAT activation in individuals with obesity and how the cold water immersions affect the BAT perfusion in humans is critical for the development of new strategies to treat obesity and its comorbidities.

DETAILED DESCRIPTION:
Obesity is a highly prevalent non-communicable disease that effects more than 20% of the population worldwide. Brown adipose tissue (BAT) has an unique ability to dissipate the energy as heat and it has been associated with metabolic benefits. Additionally, BAT has been found to be more active in young, healthy, lean individuals and to be inactive in subjects with obesity. Some studies have shown that repeated cold acclimation can enhance BAT metabolism, which is accompanied by metabolic benefits, such as improvements in insulin sensitivity. In this study we will investigate whether 12 weeks or more of cold acclimation are sufficient to improve BAT perfusion at room temperature and after 2 hours of cold exposure, and to stimulate glucose uptake (measured using 18F-FDG) in BAT after 2 hours of cold exposure. Furthermore, changes in BAT NEFA uptake will be analyzed using 18F-FTHA at room temperature. The metabolic effects of the cold acclimation protocol will be evaluated by changes in classical cardiovascular risk markers (lipid profile, glucose and insulin) after 12 weeks. Two different control groups will be included: one will include lean, healthy participants while the other will include subjects with obesity. Both groups will undergo the BAT PET/scans protocol at room temperature and after cold exposure to investigate BAT perfusion, BAT glucose uptake and BAT NEFA uptake. The volunteers with obesity will also undergo a second evaluation 12 weeks after baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30kg/m2 (for participants with obesity)
* BMI<25kg/m2 (for lean participants)
* Waist circumference >94 cm for men (for participants with obesity)
* Waist circumference > 80 for women (for participants with obesity)
* Glucose ≥7.8 and <11 mmol/L after OGTT (for participants with obesity)

Exclusion Criteria:

* Being regularly exposed to cold environments for the last 3 months (e.g. having a job as a ski monitor, fishmonger, woodcutter, etc.; or doing sports/leisure activities outdoors for prolonged periods of time, etc.)
* Having gone for winter/ice swimming and bathing more than once every 2 weeks during the last 3 months.
* Inability to undergo scanning (e.g., claustrophobia)
* Pregnancy
* Smoking (or use of nicotine based products)
* Hypo/hyperthyroidism
* Malignancies
* Immune disorders
* Viral or bacterial infections
* Abnormal cardiovascular status, arrhythmia and/or long QTc in ECG, abnormal cardiac murmur, previous history of cardiovascular disease
* Allergy to lidocaine or epinephrine, or other local anaesthetics
* Weight change (intentional or not) over the last 6-months > than 5% of body weight
* Any other cardiovascular, pulmonary, orthopaedic, neurologic, psychiatric or other conditions that in the opinion of the local clinician/researcher, would preclude participation and successful completion of the protocol, or that would negatively impact or mitigate participation in and completion of the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Brown adipose tissue perfusion | After at least 12 weeks of cold acclimation
  BAT perfusion will be measured using 15O-O2 and 15O-H2O PET-CT, at room temperature and after 2 hours of cold exposure.

SECONDARY OUTCOMES:
Brown adipose tissue glucose uptake | After at least 12 weeks of cold acclimation
  BAT glucose uptake will be measured after cold exposure using Fluorodeoxyglucose (18F-FDG).
Brown adipose tissue NEFA uptake | After at least 12 weeks of cold acclimation
  BAT NEFA uptake will be measured at room temperature using [18F]fluoro-6-thia-heptadecanoic acid (18F-FTHA).

OTHER OUTCOMES:
Metabolic parameters | After at least 12 weeks of cold acclimation
  Investigate the effects of cold acclimation on blood lipids (total, LDL and HDL cholesterol and triglycerides), fasting glucose and insulin.
Energy expenditure | After at least 12 weeks of cold acclimation
  To investigate the effects of cold acclimation on energy expenditure in fasting and postprandial states (after the intake of a mixed meal) using indirect calorimetry
BAT gene expression | After at least 12 weeks of cold acclimation
  BAT biopsies will be collected to investigate the effects of cold acclimation on BAT gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi A Virtanen, Principal Investigator — Turku University Hospital; Francisco Acosta, PhD, Study Director — Turku PET Centre; Mueez U-Din, PhD, Study Director — Turku PET Centre
Locations (1):
- Turku PET Centre, Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No